CLINICAL TRIAL: NCT02144428
Title: DETERMINATION OF HYPOALLERGENICITY TO SUBSTITUTIVE FORMULAS IN CHILDREN WITH COW'S MILK ALLERGY
Brief Title: Hypoallergenicity To Substitutive Formulas In Children With Cow's Milk Allergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: 05/14
Record Dates: First submitted 2014-05-14; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cow's milk allergy: Subjcets with a sure diagnosis of cow'a milk allergy on exclusion diet

SUMMARY:
The management of children with confirmed cow's milk allergy is based on complete avoidance of cow's milk proteins and leaves the physician with several dietary options, none of which, given the prevalence, spectrum and potential seriousness of the condition, can be recommended to all patients. In the absence of an alternative to cow's milk, the management of cow's milk allergy is based on the use of safe, affordable and nutritionally adequate formulas. Extensively hydrolyzed cow's milk protein formulas, which are considered as safe for most children with cow's milk allergy, are still liable to contain residual peptides, and hypersensitivity reactions may occur in infants allergic to cow's milk protein. Thus, specific product allergenicity must be addressed on an individual basis before recommending a formula as a substitute for cow's milk. Soy-based formula can also concomitant sensitize cow's milk allergy children to soy. Amino acid-based formulas have been studied from safety and nutritional efficacy perspectives. These formulas have been proposed for subjects highly sensitive to cow's milk protein and that cannot be managed using extensively hydolyzed formula and for children with multiple food allergies. In these conditions aminoacid based formulas are able to effectively cure allergic symptoms and to improve body growth.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a cow's milk allergy
* age between 0 to 36 months

Exclusion Criteria:

* age more than 36 months
* eosinophilic disorders of the gastrointestinal tract,
* food protein induced enterocolitic syndrome,
* concomitant chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* lactose intolerance,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal tract.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects with cow's milk allergy diagnosed by family pediatrician operating in Italy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with cow's milk allergy tolerant substitutive formulas | At diagnosis and for at least 1 months after the diagnosis
  Safety and tolerability of substitutive formulas

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy